CLINICAL TRIAL: NCT01618903
Title: A Monocenter, Open-label, Two-way Randomized Cross-over Study to Evaluate the Bioequivalence of Levetiracetam Administered as a 45 Minutes Intravenous Infusion and Same Dosage Levetiracetam Oral Tablet (Part A); and a Randomized, Double-blind, Placebo-controlled, Parallel Study on the Safety, Tolerability and Pharmacokinetics of Levetiracetam 45 Minutes Intravenous Infusion During 4 Days of b.i.d. Dosing (Part B), in Chinese Healthy Volunteers
Brief Title: An Open-label, Bioequivalence Study to Evaluate LEV Administered as a 45-min Intravenous Infusion and Same Dosage LEV Oral Tablet in Chinese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N01362A
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Human Volunteers
Keywords: Keppra Levetiracetam intravenous; Oral tablets; Bioequivalence; Pharmacokinetics; Safety; Chinese healthy volunteers
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam iv infusion (Experimental): Levetiracetam intravenous (iv) 45 min infusion administered as one single dose.
  Interventions: Drug: Levetiracetam
- Levetiracetam oral tablet (Experimental): Levetiracetam oral tablet administered as one single dose.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam 1.500 mg (500 mg/ 5 mL vials) administered as a 45 minutes intravenous infusion diluted in 100 mL 0.9 % saline solution in the morning of Day 1.
  Other Names: Keppra
  Arms: Levetiracetam iv infusion
Drug: Levetiracetam — Levetiracetam single oral administration of 3 tablets of 500 mg immediate release tablet.
  Other Names: Keppra
  Arms: Levetiracetam oral tablet

SUMMARY:
The part A of N01362 is to evaluate the bioequivalence of Levetiracetam (LEV) 1500 mg intravenous (iv) infusion when compared to tablet oral administration in Chinese healthy volunteers.

DETAILED DESCRIPTION:
The study includes 2 parts, part A is to evaluate the bioequivalence of Levetiracetam (LEV) 1500 mg intravenous (iv) infusion when compared to oral tablet, part B is to assess pharmacokinetic profile of LEV infusion during repeated dosing in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, age 18-40, weight ≥ 50 kg
* Healthy volunteers with normal vital signs, good physical and mental health status and normal electrocardiogram and laboratory test

Exclusion Criteria:

* History or presence of each systems disorders capable of altering the absorption, metabolism or elimination of drugs, or of constituting a risk factor when taking the study medication
* History or presence of drug addiction or excessive use of alcohol
* Symptomatic or asymptomatic Orthostatic Hypotension at screening
* Current smokers and former smokers
* Heavy caffeine drinker
* History of frequent and severe headache
* Any drug treatment
* Subjects who are known to have Serum Hepatitis or who are carriers of the Hepatitis B surface antigen, or Hepatitis C antibody or who are HIV positive
* Subjects on a controlled sodium diet
* Subject has made a blood donation or had a comparable blood loss

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration versus time curve from hour 0 to the time with a last quantifiable concentration (AUC(0-t)) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
Area under the plasma drug concentration-time curve from 0 to infinity (AUC) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
  The area under the curve extrapolated to infinity is calculated as the sum of AUC(0-t) and a residual part extrapolated to infinite time.
Maximum measured plasma concentration (Cmax) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
  The value of the maximum plasma concentration is directly obtained from the observed plasma concentration versus time curves.

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve calculated from 0 to 12 h (AUC(0-12)) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
Plasma concentration at the end of the 45-minutes intravenous (iv) infusion (C45'(iv)) | Pharmacokinetic samples were taken at 45 min after Levetiracetam administration
  The value of the plasma concentration at the end of the 45-min iv infusion is directly obtained from the experimental data of plasma concentration versus time curves.
Time to reach the maximum plasma concentration of Levetiracetam after administration (tmax) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
Terminal half-life of Levetiracetam (t1/2) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
  The terminal half-life associated with the terminal rate constant λ_z is calculated as: ln2/λ_z. λ_z is the first order rate constant of elimination.
Total body clearance after intravenous infusion of Levetiracetam (CL(iv)) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
  The CL(iv) is calculated as:
  CL=Dose of LEV/AUC.
Apparent total body clearance after oral administration of Levetiracetam (CL/F(tablet)) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
  The CL/F (tablet) is calculated as:
  CL/F=Dose of LEV/AUC.
Volume of distribution after intravenous infusion of Levetiracetam (Vz(iv)) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
  The volume of distribution after iv infusion is calculated as:
  Vz=CL/λ_z, where CL is the total body clearance and λ_z the first order rate constant of elimination.
Apparent volume of distribution after oral administration of Levetiracetam (Vz/F(tablet)) | Pharmacokinetic samples were taken from pre-dose to 36 hours after Levetiracetam administration
  The apparent volume of distribution after oral administration is calculated as:
  Vz/F= (CL/F)/λ_z.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Shanghai, China

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm